CLINICAL TRIAL: NCT07081906
Title: A Prospective and Randomized Study of Efficacy and Safety of Transdermal Oxybutynin Versus Oral Oxybutynin in The Management of Children With Overactive Bladder
Brief Title: Transdermal Versus Oral Oxybutynin in Pediatric OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Halil Sevinc, MD - Urology Specialist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kartalcity_ahs_01
Record Dates: First submitted 2025-07-09; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Overactive Bladder (OAB); Drug Delivery Systems; Anticholinergic Side Effects; Children and Adolescents, Boys and Girls
Keywords: overactive bladder; oxybutynin; transdermal; children; anticholinergic side effects
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — oxybutynin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Oxybutynin (Active Comparator): Participants received oral oxybutynin suspension (5 mg, 2-3 times daily depending on body weight) for 3 months.
  Interventions: Drug: Oral Oxybutynin
- Transdermal oxybutynin (Active Comparator): Participants received transdermal oxybutynin patch (3.9 mg/day) applied twice weekly for 3 months.
  Interventions: Drug: transdermal oxybutinin

INTERVENTIONS:
Drug: Oral Oxybutynin — The oral form of oxybutinin was preferred for patients who had no difficulty swallowing and whose families preferred a conventional administration route. Medication was given under parental supervision to ensure adherence. Patients were monitored monthly for potential anticholinergic side effects. The patch form of oxybutinin was chosen for patients who experienced difficulties with oral intake or had previous intolerance to oral anticholinergics. Application sites were rotated to reduce the risk of local skin reactions. Families received instructions on proper patch application technique.
  Arms: Oral Oxybutynin
Drug: transdermal oxybutinin — The oral form of oxybutinin was preferred for patients who had no difficulty swallowing and whose families preferred a conventional administration route. Medication was given under parental supervision to ensure adherence. Patients were monitored monthly for potential anticholinergic side effects. The patch form of oxybutinin was chosen for patients who experienced difficulties with oral intake or had previous intolerance to oral anticholinergics. Application sites were rotated to reduce the risk of local skin reactions. Families received instructions on proper patch application technique.
  Arms: Transdermal oxybutynin

SUMMARY:
This is a prospective, randomized controlled clinical trial designed to compare the efficacy and safety of transdermal versus oral oxybutynin in children diagnosed with overactive bladder (OAB) who remain symptomatic despite conservative management. A total of 90 children were planned to be enrolled and randomized to receive either oral oxybutynin suspension or a transdermal oxybutynin patch. The primary outcome was defined as the change in Dysfunctional Voiding and Incontinence Symptom Score (DVISS) from baseline to the end of the treatment period. Secondary outcomes included changes in urinary frequency, voided volume, maximum flow rate (Qmax), and the incidence of adverse events. The study aimed to assess whether the transdermal route of administration provides an alternative therapeutic option with favorable tolerability in pediatric OAB patients.

ELIGIBILITY:
Inclusion Criteria:

* Persistent symptoms of overactive bladder (OAB) despite at least 3 months of conservative treatment (e.g., behavioral therapy, planned fluid intake, and voiding schedules)
* No prior medical or surgical treatment for OAB
* Ability to attend follow-up visits with family/guardian
* Written informed consent obtained from a legal guardian

Exclusion Criteria:

* History of febrile or recurrent urinary tract infections
* Presence of urethral stricture
* Known or suspected neurogenic bladder dysfunction
* Previous bladder surgery
* History of urolithiasis (kidney stones)
* Contraindications to oxybutynin therapy

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Dysfunctional Voiding and Incontinence Symptom Score (DVISS) | From enrollment to the end of treatment at three months
  The primary outcome was the change in DVISS score, a validated questionnaire assessing lower urinary tract symptoms in children. Scores range from 0 to 35, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet H Sevinc, MD, Urology Specialist, Principal Investigator — Kartal Dr. Lütfi Kırdar Training and Research Hospital
Locations (1):
- Kartal Dr. Lütfi Kırdar Training and Research Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No